CLINICAL TRIAL: NCT04199260
Title: Investigación clínica Para la evaluación Del Efecto de PAPILOCARE® en la normalización de Las Alteraciones citológicas Del Cuello Del útero Causadas Por el VPH
Brief Title: Investigation to Evaluate PAPILOCARE® Gel Effect on Normalization of Cervix Cytological Alterations Caused by HPV.
Acronym: PAPILOBS
Status: Completed | Type: Observational
Sponsor: Procare Health Iberia S.L. (Industry)
Collaborators: Adknoma Health Research (Industry)
Responsible Party: Sponsor
Other Study IDs: PAPILOBS-2017-01
Record Dates: First submitted 2019-12-11; First posted 2019-12-13 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: HPV Infection; Lesion Cervix
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Papilocare: all patients gonna received papilocare treatment as per usual practice.
  Interventions: Device: papilocare vaginal gel

INTERVENTIONS:
Device: papilocare vaginal gel — Papilocare is a gel vaginally administered by a single-dose cannula. Vaginal gel formulation is effective as a local treatment with controlled systemic absorption and rapid and efficient distribution

SUMMARY:
Observational clinical study, national, multicentric, prospective, non-comparative, with medical device, under application consistent with CE marking, for the evaluation of Papilocare® effectivness in the normalization of cervix cytological abnormalities caused by HPV.

DETAILED DESCRIPTION:
300 patients will be included in approximately 50 Spanish sites. The study comprehend a maximum of 3 visits. At visit 1, patient's writted informed consent will be collected, patient's selection critera will be checked, and patient's medial history data will be collected. At visit 2, 6 months after the first visit, the primary and secondary objectives will be evaluated. For those patients who finish treatment after 6 months, this will be the final visit. Only in that cases where, by usual clinical practice, the doctor indicates patient should continue under treatment, visit 3, wich will take place 12 months after streatment stars, will be the last visit for the patient under study.

ELIGIBILITY:
Inclusion Criteria:

1. Woman over 25 years, whether or not they have been vaccinated against HPV.
2. Able to read and understand the Patient Information Sheet and the Informed Consent form and accept the participation in the study by signing the Informed Consent form.
3. Patient who comes to a visit with a routine cytological result of ASCUS or LSIL and HPV-positive test, of at most 3 months prior to the start of treatment with Papilocare®.
4. Patient who, under that situation, undergoes a colposcopy and has a concordant result with cytology.
5. Patient who has been prescribed treatment with Papilocare® by medical decision prior to their participation in the study.

Exclusion Criteria:

1. Any situation / alteration / pathology, gynecological or not, which, in medical judgment, does not advise or contraindicate the use of Papilocare®.
2. Women of childbearing age who do not use effective contraceptive methods, pregnant women, suspected pregnancy, desire for the same within the next 6 months or during breastfeeding.
3. Participation in any one clinical trial at present or in the 4 weeks prior to inclusion in the study.
4. Any planned surgery that precludes correct compliance with the guideline.
5. Known allergies to any of the components of Papilocare®.

Min Age: 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The main objective of the study is to evaluate the degree of normalization of cytological abnormalities of the cervix caused by HPV. For this purpose, women over 25 years old with positive HPV with lesions in the cervical mucosa, and concordant colposcopic image have been chosen as the target population.
  No exceptional measures are planned for the recruitment of patients in this study.
Sampling Method: Probability Sample
Enrollment: 263 (Actual)
Dates: Start 2018-05-20 (Actual); Primary Completion 2021-02-18 (Actual); Study Completion 2021-02-18 (Actual)

PRIMARY OUTCOMES:
Percentage of patient who normalized their cytology with concordant colposcopy. | 6 months
  The percentage of patients with normalization of the cytology with concordant colposcopy, at 6 months, and at 12 months if applicable, has been established as the main variable of the study, in order to assess the degree of normalization of cytological alterations.
  Colposcopy concordant with normalized cytology results will be considered those colposcopic findings classified as normal, non-specific or as abnormal grade 1 (minor) according to the definition of the Nomenclature Committee of the International Federation of Cervical and Colposcopic Pathology (IFCPC). accepted at the Rio World Congress, July 5, 2011.
Percentage of patient who normalized their cytology with concordant colposcopy. | 12 months if applicable
  The percentage of patients with normalization of the cytology with concordant colposcopy, at 6 months, and at 12 months if applicable, has been established as the main variable of the study, in order to assess the degree of normalization of cytological alterations.
  Colposcopy concordant with normalized cytology results will be considered those colposcopic findings classified as normal, non-specific or as abnormal grade 1 (minor) according to the definition of the Nomenclature Committee of the International Federation of Cervical and Colposcopic Pathology (IFCPC). accepted at the Rio World Congress, July 5, 2011.

SECONDARY OUTCOMES:
Percentage of patient who clear partially or completely the presence of HPV | 6 months
  To evaluate the clearance of HPV, the percentage of patients with total or partial clearance of HPV measured by PCR or genetic diagnostic kits that allow the identification of strains at 6 months (and 12 months if applicable) from the start of treatment.
Percentage of patient who clear partially or completely the presence of HPV | 12 months if applicable
  To evaluate the clearance of HPV, the percentage of patients with total or partial clearance of HPV measured by PCR or genetic diagnostic kits that allow the identification of strains at 6 months (and 12 months if applicable) from the start of treatment.
Patient's satisfaction degree with the study treatment | 6 months
  Changes appreciated in the Likert scale at 6 months (and at 12 months if applicable) of the start of treatment will be used to evaluate satisfaction degree with the use of Papilocare gel as treatment.
Patient's satisfaction degree with the study treatment | 12 months if applicable
  Changes appreciated in the Likert scale at 6 months (and at 12 months if applicable) of the start of treatment will be used to evaluate satisfaction degree with the use of Papilocare gel as treatment.
Safety and tolerability of treatment | 6 months
  The incidence, nature and severity of adverse events during the 6 months (or 12 months if applicable) of the duration of the treatment will be used to assess the safety and tolerability of treatment.
Safety and tolerability of treatment | 12 months if applicable
  The incidence, nature and severity of adverse events during the 6 months (or 12 months if applicable) of the duration of the treatment will be used to assess the safety and tolerability of treatment.

OTHER OUTCOMES:
Evaluate the results of the biopsy (optional) | 6 months
  To assess the effect on biopsies (when available), the percentage of patients who improve and those who maintain the degree of histological alteration have been established at 6 months (and at 12 months if applicable) of the start of treatment.
Evaluate the results of the biopsy (optional) | 12 months if applicable
  To assess the effect on biopsies (when available), the percentage of patients who improve and those who maintain the degree of histological alteration have been established at 6 months (and at 12 months if applicable) of the start of treatment.

CONTACTS AND LOCATIONS:
Locations (9):
- Spain (9):
  - Hospital General Universitario de Alicante, Alicante
  - Women´s Health Institute, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Clínica Diatros, Barcelona
  - Gabinete Médico Velázquez, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Instituto Palacios de Salud y Medicina de la Mujer, Madrid
  - MD Anderson, Madrid
  - Hospital Quirón Málaga, Málaga

IPD SHARING:
Plan to Share IPD: Undecided